CLINICAL TRIAL: NCT07282938
Title: Combined Effects of Soft Robotic Hand and Electrical Stimulation on Hand Function in Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/040 Amna
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Cerebro-vascular Accident
Keywords: Stroke; hand impairments; soft robotic hand; electrical stimulation; robotic therapy; Cerebrovascular accident
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: After recruitment, the participants will be allocated into their respective groups utilizing the online randomizer tool.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded study approach will be utilized. Participants and outcome assessor both will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group-1 (Soft Robotic Hand + Neuromuscular Electrical Stimulation) (Experimental): The experimental group will follow a rehabilitation program that combines soft robotic hand support along with electrical muscle stimulation (EMS), and perform task oriented training. Syrebo Hand rehabilitation robotic glove will be used which help the patient to flex and extend the fingers as in open or close a fist and for the stimulation of muscles ComfyStim EMS device will be used, By placing EMS electrodes on the important muscle groups used for gripping, moving the wrist, and making small movements, adjusting the intensity to what each person can handle. After the careful set up of both devices patient will perform task training such as grip-release cycles, reaching to grab objects, pinching small items, and mimicking daily activities like lifting a cup or stacking blocks.
  Interventions: Other: Soft Robotic Hand combined with Neuromuscular Electrical Stimulation along with Task Oriented Training
- Control: Group-2 ( Neuromuscular Electrical Stimulation) (Other): The control group will follow a rehabilitation program that combines support of electrical stimulation, and task oriented training. For the stimulation of muscles ComfyStim EMS device will be used, by placing EMS electrodes on the important muscle groups used for gripping, moving the wrist, and making small movements, adjusting the intensity to what each person can handle. After the careful set up of EMS device patient will perform task training such as grip-release cycles, reaching to grab objects, pinching small items, and mimicking daily activities like lifting a cup or stacking blocks.
  Interventions: Other: Neuromuscular Electrical Stimulation along with Task Oriented Training

INTERVENTIONS:
Other: Soft Robotic Hand combined with Neuromuscular Electrical Stimulation along with Task Oriented Training — Group-1, will follow a rehabilitation program that combines soft robotic hand support, electrical muscle stimulation (EMS), and task oriented training. After the adjustment of soft robotic hand, EMS electrodes will be placed on specific muscles, with set FITT principal as, A pulse frequency of 20 to 50 Hz and a pulse duration of 400 μs will be set with the intensity as per tolerated by the participant. Participants will perform task oriented activities that will include, Reaching to grasp objects, Picking up and releasing things at different heights using active finger and wrist extension. Opening a jar, or bottle, Turning a key or doorknob, Holding and lifting a tray or flat object, Pushing objects forward (like sliding a book across) with the assistance of soft robotic hand while electrical simulations are being delivered through the EMS for 40 min/day, 03 days/week, for 08 week. Measurements will be taken prior to the treatment, after 4 weeks of treatment and 8 weeks post-treatment.
  Other Names: Soft Robotic Hand; robotic assisted therapy; electrical stimulation; soft robotic hand and electrical stimulation; task oriented training
  Arms: Experimental: Group-1 (Soft Robotic Hand + Neuromuscular Electrical Stimulation)
Other: Neuromuscular Electrical Stimulation along with Task Oriented Training — The control group will follow a rehabilitation program that combines support of electrical stimulation, and task oriented training. For the stimulation of muscles ComfyStim EMS device will be used. The FITT principal used for EMS will be as, A pulse frequency of 20 to 50 Hz and a pulse duration of 400 μs will be set with the intensity as per tolerated by the participant. Participants will perform task oriented activities that will include, Reaching to grasp objects, Picking up and releasing things at different heights using active finger and wrist extension. Opening a jar or bottle, Turning a key or doorknob, Holding and lifting a tray or flat object, Pushing objects forward (like sliding a book across) while electrical simulations are being delivered through the EMS for 40 min/day, 03 days/week, for 08 week. Measurements will be taken prior to the treatment, after 4 weeks of treatment and 8 weeks post-treatment.
  Other Names: Electrical stimulation; Neuromuscular electrical stimulation; task oriented training
  Arms: Control: Group-2 ( Neuromuscular Electrical Stimulation)

SUMMARY:
Stroke is a clinically delineated syndrome, which is characterised by an acute, focal neurological deficit resulting from vascular injury (infarction or haemorrhage) within the central nervous system. Notably, around 80 percent of stroke survivors experience post-stroke deficits in upper extremity (UE) motor performance, impacting grip strength, dexterity, and functional independence, which greatly hinder the ability of stroke patients to carry out activities of daily living (ADL), and in turn affects their overall quality of life (QOL).One potential solution to these difficulties is the creation of rehabilitation robotic devices that incorporate hand technology and electrical stimulation. Although soft robotic assistive devices and electrical stimulation have each shown positive effects on motor recovery, their combined use has yet to be thoroughly investigated. This study intends to determine if the simultaneous application of these therapies can speed up rehabilitation results in comparison to independent therapies. Stroke Participants will be divided into two groups, Experimental group and Control group. Both the groups will receive intervention for 40 min/day, 03 days/week, for 08 week and measurements will be taken prior to the treatment, after 4 weeks of treatment and 8 weeks post-treatment.

DETAILED DESCRIPTION:
Stroke is the second largest cause of death and disability worldwide. On the basis of cause, there are two major kinds of strokes, 80 % of which are ischemic strokes and 20% are of hemorrhagic stroke. While on the basis of duration stroke is divided as transient ischemic stroke (TIA), acute, sub-acute and chronic stroke. Between 1993/1994 and 2005, the mean age of stroke onset decreased by two years, and the proportion of strokes among individuals aged 20 to 54 increased by approximately 50%, from 12.9% to 18.6%, with ischemic stroke being the most common type. Prevalence of stroke in low-income countries is increasing over the last three decades with an annual increase of 14.3%, and globally, the overall prevalence of stroke in the elderly is estimated at 7.4%. Between 17% and 40% of stroke survivors experience spasticity in their upper extremities, significantly impairing their ability to perform daily tasks. Rehabilitation of the upper limbs is particularly crucial during the first six months following a stroke, as recovery of motor functions and daily living activities significantly diminishes after this period. Beyond this six-month window, up to 66% of patients fail to regain functional upper-limb capabilities. Robot assisted therapy (RAT) is a novel approach used in the stroke rehabilitation to deliver the motor and task-oriented training by utilizing robotic devices. There are many researches working on the effect of soft robotic hand and electrical stimulation and their effect compared with the other physical therapy intervention that are constrained induced movement therapy (CIMT) or Mirror therapy or traditional physical therapy program, but the results for the combined effect of the soft robotic hand and electrical stimulation when applied along with functional task training are still under study. Given the limitations of traditional therapies, the integration of soft robotic hand with electrical stimulation may offer a promising approach to early rehabilitation. This integrated approach can enhance functional recovery by facilitating neuroplasticity and motor relearning through synchronised passive and active movements, thereby promoting greater independence in daily activities. This research aims to develop effective rehabilitation strategies that lower long-term healthcare costs and enhance overall motor recovery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with their first episode of stroke.
* Participants with 3-6 months post stroke.
* Participants with normal cognition on Montreal Cognitive Assessment (MOCA) ≥24.
* Participants with the ability to extend Metacarpophalangeal (MCP) and Proximal Interphalangeal (PIP) joint to 180 degree passively
* Modified Ashworth Scale < 2.
* Participants with the score of 10 to 16 on National Institute of Health Stroke Scale Score (NIHSS Score).

Exclusion Criteria:

* Presence of other neurological, neuromuscular, orthopedic diseases, or
* conditions that may interfere with task performance.
* Participants with sensory disturbances in the fingers

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test | Measurements will be taken before the treatment as baseline, after 4 weeks of treatment, and 8 weeks post-treatment
  Motor hand function will be assessed using the Wolf Motor Function Test (WMFT). The WMFT evaluates functional ability and movement speed through 17 tasks, including 15 timed functional tasks and 2 strength-based tasks. Each task is scored on a 6-point scale (0-5), with higher scores indicating better performance; total scores range from 0 to 85.
Fugl-meyer assessment of upper limb (FMA-UE) | Measurements will be taken before the treatment, after 4 weeks of treatment, and 8 weeks post-treatment
  Motor hand function will be assessed using the Fugl-Meyer Assessment of Upper Extremity (FMA-UE). The FMA-UE has demonstrated excellent test-retest and inter- and intra-rater reliability, and evidence for its content validity. The FMA assesses motor recovery in the upper extremity using a 33-item scale scored from 0 to 2 per item, with a maximum score of 66.
Nine-Peg Hole Test | Measurements will be taken before the treatment, after 4 weeks of treatment, and 8 weeks post-treatment
  Dexterity of the affected hand will be assessed using the Nine-Hole Peg Test (NHPT), a standardized and widely used tool for measuring fine motor coordination. Participants are instructed to place nine pegs into nine holes on a board and then remove them as quickly as possible, using one hand at a time. The total time taken to complete the task is recorded in seconds. Shorter completion times indicate better manual dexterity.
Dynamometer | Measurements will be taken before the treatment, after 4 weeks of treatment, and 8 weeks post-treatment
  Grip strength will be assessed using a hand-held dynamometer, a reliable tool for measuring isometric muscle force. Participants will be instructed to squeeze the device with maximum effort while seated, with the elbow flexed at 90 degrees and the forearm in a neutral position. Each hand will be tested three times, and the highest value will be recorded. This method provides an objective measure of hand strength and is commonly used in stroke rehabilitation to monitor functional recovery and response to intervention.
Modified Ashworth Scale | Measurements will be taken before the treatment, after 4 weeks of treatment, and 8 weeks post-treatment.
  The Modified Ashworth Scale (MAS) will be used to evaluate muscle spasticity in the affected upper limb. This scale grades resistance during passive soft-tissue stretching on a 6-point ordinal scale (0 to 4, with an additional 1+ grade), where higher scores indicate increased muscle tone. MAS is widely used in stroke rehabilitation to monitor changes in spasticity and assess the effectiveness of interventions aimed at promoting motor recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Lahore University of Biological and Applied sciences, UBAS
Locations (2):
- Pakistan (2):
  - Pakistan Society for the Rehabilitation of the Disabled (PSRD), Lahore, Punjab Province
  - Shadman Medical Center, Stroke Rehabilitation, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kristensen MGH, Busk H, Wienecke T. Neuromuscular Electrical Stimulation Improves Activities of Daily Living Post Stroke: A Systematic Review and Meta-analysis. Arch Rehabil Res Clin Transl. 2021 Nov 12;4(1):100167. doi: 10.1016/j.arrct.2021.100167. eCollection 2022 Mar. PMID 35282150
- [Background] Ko MJ, Chuang YC, Ou-Yang LJ, Cheng YY, Tsai YL, Lee YC. The Application of Soft Robotic Gloves in Stroke Patients: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Brain Sci. 2023 Jun 2;13(6):900. doi: 10.3390/brainsci13060900. PMID 37371378
- [Background] Bayindir O, Akyuz G, Sekban N. The effect of adding robot-assisted hand rehabilitation to conventional rehabilitation program following stroke: A randomized-controlled study. Turk J Phys Med Rehabil. 2022 Jun 1;68(2):254-261. doi: 10.5606/tftrd.2022.8705. eCollection 2022 Jun. PMID 35989963
- [Background] Chen P, Liu TW, Tse MMY, Lai CKY, Tsoh J, Ng SSM. The Predictive Role of Hand Section of Fugl-Meyer Assessment and Motor Activity Log in Action Research Arm Test in People With Stroke. Front Neurol. 2022 Jul 7;13:926130. doi: 10.3389/fneur.2022.926130. eCollection 2022. PMID 35873769
- [Background] Chien WT, Chong YY, Tse MK, Chien CW, Cheng HY. Robot-assisted therapy for upper-limb rehabilitation in subacute stroke patients: A systematic review and meta-analysis. Brain Behav. 2020 Aug;10(8):e01742. doi: 10.1002/brb3.1742. Epub 2020 Jun 26. PMID 32592282
- [Background] Lindsay LR, Thompson DA, O'Dell MW. Updated Approach to Stroke Rehabilitation. Med Clin North Am. 2020 Mar;104(2):199-211. doi: 10.1016/j.mcna.2019.11.002. PMID 32035564
- [Background] Mosconi MG, Paciaroni M. Treatments in Ischemic Stroke: Current and Future. Eur Neurol. 2022;85(5):349-366. doi: 10.1159/000525822. Epub 2022 Aug 2. PMID 35917794
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228